CLINICAL TRIAL: NCT02819375
Title: Inonu University Faculty of Medicine Department of Anesthesiology and Reanimation
Brief Title: Comparison of Propofol, Propofol-remifentanil and Propofol-ketamine Anesthesia During Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ulku 2
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Electroconvulsive Therapy
Keywords: propofol; ketamine; remifentanil
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Propofol (Active Comparator): anesthesia will induced 1 mg/kg propofol
  Interventions: Drug: Propofol
- Group propofol/remifentanil (Active Comparator): anesthesia will induced 0.5 mg/kg propofol and 1 µg/kg remifentanil
  Interventions: Drug: Propofol+Remifentanil
- Group propofol/ketamine (Active Comparator): anesthesia will induced propofol 0.5 mg/kg and ketamine 0.5 mg/kg
  Interventions: Drug: Propofol+Ketamine

INTERVENTIONS:
Drug: Propofol — 1 mg/kg propofol
  Other Names: Diprivan
  Arms: Group Propofol
Drug: Propofol+Remifentanil — 0.5 mg/kg propofol+0.5 mg/kg remifentanil
  Other Names: Propofol+Ultiva
  Arms: Group propofol/remifentanil
Drug: Propofol+Ketamine — 0.5 mg/kg propofol and 0.5 mg/kg ketamine
  Other Names: Propofol+Ketalar
  Arms: Group propofol/ketamine

SUMMARY:
Electroconvulsive therapy (ECT) is a common treatment method used in severe depression and other psychiatric diseases. Currently, most ECT procedures are carried out with muscle paralysis under general anaesthesia. The anticonvulsant properties of sedative and hypnotic drugs used during general anaesthesia may reduce the efficacy of ECT. It is important to establish an accurate balance between adequate anaesthesia depth and optimal seizure duration.

We aimed to compare the effectiveness of three anaesthetic regimens (propofol alone, propofol with remifentanil and propofol with ketamine), with respect to seizure duration and seizure quality in patients undergoing electroconvulsive therapy.

DETAILED DESCRIPTION:
In this study, 45 patients of American Society of Anesthesiologists (ASA) physical status I-II aged between 18-60 years who were scheduled for ECT sessions under general anesthesia. Seven consecutive ECT sessions will evaluated in this study. Exclusion criteria; pregnancy, cerebrovascular disease, epilepsy, unstable cardiovascular disease, chronic obstructive pulmonary disease, and renal or hepatic failure.

Electrocardiogram (ECG), noninvasive arterial blood pressure, and peripheral oxygen saturation (SpO2) measurements will utilized along with standard monitoring techniques in the operating room for patients who did not receive pre-operative medication. A 20-gauge intravenous cannula will placed before induction of patients. Each patient will receive either propofol 1 mg/kg alone (Group P), propofol 0.5 mg/kg and remifentanil 1 µg/kg (Group R), or propofol 0.5 mg/kg and ketamine 0.5 mg/kg (Group K) for their all electroconvulsive therapy session. A pneumatic tourniquet will applied to the arm and then will inflated to isolate blood circulation and allow for an accurate assessment of the motor seizure. Rocuronium (0.3 mg/kg bolus) will administered intravenously and ventilation will assisted using a facemask and 100% oxygen in three groups. Electrostimulus will performed via bifrontotemporal electrodes with a Thymatron System IV ECT Instrument (Somatics Inc.; Lake Bluff, IL, USA) by a psychiatrist who was blind to the study groups. In the initial session, patients will received ECT with 30-50% of the maximum output stimulus, depending on the preference of the psychiatrist. Thereafter, the same psychiatrist will arranged the stimulus amplitudes according to the clinical results of each patient.

The duration of the EEG, motor seizure, and postictal suppression index (PSI) will recorded from the EEG and electromyography traces. Heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), and peripheral oxygen saturation (SpO2) values will taken before anesthesia induction (Tbaseline), after the induction (T0), and following the ECT session at 1 (T1), 3 (T3), and 10 (T10) minutes. Time from the end of rocuronium administration to the time of recovery of spontaneous breathing, time of eye opening, and time of obeying verbal commands will recorded. The presence of complications, such as arrhythmia, laryngospasm, and agitation, will also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Study include 45 patients of American Society of Anesthesiologists (ASA) physical status I-II aged between 18-60 years who scheduled for ECT sessions under general anesthesia

Exclusion Criteria:

* Pregnancy
* Cerebrovascular disease
* Epilepsy
* Unstable cardiovascular disease
* Chronic obstructive pulmonary disease
* Renal or hepatic failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
seizure activity | intraoperative
  Motor (EMG) and electroencephalogram (EEG) seizure durations

SECONDARY OUTCOMES:
heart rate (HR) | (approximately 10 minutes for all measurements) prior to the seizure, after the anesthetic induction, and following the ECT session at 1 minute, 3 minutes, and 10 minutes
  heart rate
mean arterial pressure (MAP) | (approximately 10 minutes for all measurements) prior to the seizure, after the anesthetic induction, and following the ECT session at 1 minute, 3 minutes, and 10 minutes
  mean arterial pressure
recovery times | intraoperative
  Recovery times will be assessed with spontaneous breathing, eye opening, obeying

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Ozgul, Ass.Prof., Principal Investigator — Inonu University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erdogan Kayhan G, Yucel A, Colak YZ, Ozgul U, Yologlu S, Karlidag R, Ersoy MO. Ketofol (mixture of ketamine and propofol) administration in electroconvulsive therapy. Anaesth Intensive Care. 2012 Mar;40(2):305-10. doi: 10.1177/0310057X1204000214. PMID 22417026
- [Result] Begec Z, Erdogan Kayhan G, Toprak HI, Sahin T, Konur H, Colak C, Durmus M, Ersoy MO. Sevoflurane alone and propofol with or without remifentanil for electroconvulsive therapy-a randomised, crossover study. Anaesth Intensive Care. 2013 Mar;41(2):202-6. doi: 10.1177/0310057X1304100209. PMID 23530786